CLINICAL TRIAL: NCT05632302
Title: A Pilot Study to Estimate Intracranial Pressure Noninvasively in Traumatic Brain Injury Patients
Brief Title: A Non-invasive Intracranial Pressure (nICP) Monitoring System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Crainio Ltda (Industry)
Collaborators: City, University of London (Other); Barts & The London NHS Trust (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 219476
Record Dates: First submitted 2022-11-11; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Traumatic Brain Injury; Intracranial Hypertension
Keywords: Intracranial pressure; Near infrared spectroscopy; Photoplethysmography; Noninvasive monitoring
MeSH Terms: conditions — Brain Injuries, Traumatic; Intracranial Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TBI-ICP monitoring (Experimental): Optical signals acquisition from the nICP probe stuck to the patient's forehead
  Interventions: Device: nICP

INTERVENTIONS:
Device: nICP — The nICP probe contains infrared light sources that illuminate the deep brain tissue of the frontal lobe. Photodetectors in the probe detect the backscattered light, which is modulated by pulsation of the cerebral arteries.

SUMMARY:
Researchers have developed a probe that contains infrared light sources that can illuminate the deep brain tissue of the frontal lobe. Photodetectors in the probe detect the backscattered light, which is modulated by pulsation of the cerebral arteries. Changes in the extramural arterial pressure affect the morphology of the recorded optical pulse, so analysis of the acquired signal using an appropriate algorithm could enable the calculation of the intracranial pressure noninvasively (nICP), which would be displayed to clinicians continuously.

This pilot study is the first evaluation of the device in patients in who the gold standard comparator of invasive ICP was available. The acquisition of pulsatile optical signals was performed for up to 48 hours in each of the 40 patients who were undergoing invasive ICP monitoring as part of their normal medical treatment.

Features of the optical signals would be analysed offline. A machine vector support algorithm would be implemented, with the aim of estimating ICP noninvasively and compared to the gold standard of synchronously acquired invasive ICP data.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is the most common cause of death and disability in the under 40 age group both in the United Kingdom and worldwide, and prevalence is increasing. The mainstay of severe TBI management is intracranial pressure (ICP) measurement. ICP is defined as the pressure within the skull and brain. TBI often causes a rise in ICP as the brain swells within the rigid skull and therapy is directed at keeping this pressure at an acceptable level with medications or surgery. Very high ICP may lead to further brain damage resulting in increased disability or death.

Existing techniques to measure ICP involve placing an electrical sensor into the brain tissue through a small hole drilled in the skull. This procedure risks infection and bleeding into the brain and can only be performed by a neurosurgeon. Therefore, there is a vital demand to develop non-invasive technologies that will allow measuring the ICP without inserting a sensor in the brain. This technology will decrease the risks, permit monitoring outside the hospital (eg in an ambulance) and reduce the costs. It will also increase the indication for ICP monitoring to include other conditions (e.g. stroke or brain tumours) which are not currently monitored.

The proposed non-invasive ICP (nICP) monitor works by shining a harmless light into the brain through the skull. The developed sensor was attached to the skin of the forehead and recorded optical signals (known as photoplethysmography (PPG)) from the brain, which are related to changes in the ICP. This pilot aims to build the first clinical database of nICP signals in intensive care patients. The acquisition of an extensive set of signals would allow the generation of advanced algorithms and Machine Learning (ML) models utilising optical signal feature extraction techniques. The resulting model will be implemented in translating the optical signals into absolute measurements of ICP.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to the Royal London Hospital who is having invasive ICP monitoring as part of their normal medical care
* Subject is able to understand the risks and potential benefits of participating in the study and is willing to provide written informed consent. If the patient is unconscious, and a consultee is not available then a professional consultee (a doctor looking after the patient who is not involved in the trial) will assent to inclusion in the trial and non-invasive ICP monitoring will be performed.

Exclusion Criteria:

* Patients with decompressive craniectomy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Machine learning model agreement | 48 hours record per patient
  Bland-Altman limits of agreement between the offline estimation of nICP and the invasive ICP measurements

SECONDARY OUTCOMES:
Machine learning model diagnostic accuracy | 48 hours record per patient
  Sensitivity and specificity of the offline nICP estimation to identify ICP values over 20 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Uff, FRCS, Principal Investigator — Consultant Neurosurgeon (Royal London Hosptial)
Locations (1):
- Royal London Hospital, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Only the final results of the nICP safety and accuracy would be published. Any individual participant data would be available to other researchers.

REFERENCES:
- [Background] Head injury: assessment and early management. London: National Institute for Health and Care Excellence (NICE); 2019 Sep. Available from http://www.ncbi.nlm.nih.gov/books/NBK552670/ PMID 31944644
- [Background] Lawrence T, Helmy A, Bouamra O, Woodford M, Lecky F, Hutchinson PJ. Traumatic brain injury in England and Wales: prospective audit of epidemiology, complications and standardised mortality. BMJ Open. 2016 Nov 24;6(11):e012197. doi: 10.1136/bmjopen-2016-012197. PMID 27884843
- [Background] Raboel PH, Bartek J Jr, Andresen M, Bellander BM, Romner B. Intracranial Pressure Monitoring: Invasive versus Non-Invasive Methods-A Review. Crit Care Res Pract. 2012;2012:950393. doi: 10.1155/2012/950393. Epub 2012 Jun 8. PMID 22720148
- [Background] Kawoos U, McCarron RM, Auker CR, Chavko M. Advances in Intracranial Pressure Monitoring and Its Significance in Managing Traumatic Brain Injury. Int J Mol Sci. 2015 Dec 4;16(12):28979-97. doi: 10.3390/ijms161226146. PMID 26690122
- [Background] Nag DS, Sahu S, Swain A, Kant S. Intracranial pressure monitoring: Gold standard and recent innovations. World J Clin Cases. 2019 Jul 6;7(13):1535-1553. doi: 10.12998/wjcc.v7.i13.1535. PMID 31367614
- [Background] Roldan M, Chatterjee S, Kyriacou PA. Brain Light-Tissue Interaction Modelling: Towards a non-invasive sensor for Traumatic Brain Injury. Annu Int Conf IEEE Eng Med Biol Soc. 2021 Nov;2021:1292-1296. doi: 10.1109/EMBC46164.2021.9630909. PMID 34891522
- [Background] Roldan M, Kyriacou PA. Near-Infrared Spectroscopy (NIRS) in Traumatic Brain Injury (TBI). Sensors (Basel). 2021 Feb 24;21(5):1586. doi: 10.3390/s21051586. PMID 33668311
- [Background] Roldan M, Abay TY, Kyriacou PA. Non-Invasive Techniques for Multimodal Monitoring in Traumatic Brain Injury: Systematic Review and Meta-Analysis. J Neurotrauma. 2020 Dec 1;37(23):2445-2453. doi: 10.1089/neu.2020.7266. Epub 2020 Sep 24. PMID 32821023
- [Derived] Roldan M, Abay TY, Uff C, Kyriacou PA. A pilot clinical study to estimate intracranial pressure utilising cerebral photoplethysmograms in traumatic brain injury patients. Acta Neurochir (Wien). 2024 Feb 27;166(1):109. doi: 10.1007/s00701-024-06002-4. PMID 38409283